CLINICAL TRIAL: NCT07303556
Title: Improving the Diagnosis and Treatment of Cardiovascular Diseases in Kazakhstan by Introducing Correction of Metabolism With Glucagon-like Peptide 1 (GLP-1) Drugs
Brief Title: Improving Cardiovascular Disease Diagnosis and Treatment in Kazakhstan Using Metabolic Correction With GLP-1 Drugs
Acronym: ICDDTKZ26
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazarbayev University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BR24993023
Record Dates: First submitted 2025-07-30; First posted 2025-12-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Diabete Type 2; Arterial Hypertension
Keywords: Heart Failure; Diabete Type 2; Preserved Ejection Fraction; Sequencing
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Hypertension | interventions — Tirzepatide; dapagliflozin; empagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients with heart failure and preserved ejection fraction (EF ≥ 45%) (Experimental): Participants diagnosed with chronic heart failure with preserved ejection fraction (EF ≥ 45%) who receive treatment with glucagon-like peptide-1 (GLP-1) receptor agonists
  Interventions: Drug: Tirzepatide (Mounjaro); Drug: dapagliflozin, empagliflozin, metformin
- Patients with chronic heart failure with preserved ejection fraction (EF ≥ 45%) and type 2 diabetes (Experimental): Participants diagnosed with heart failure with preserved ejection fraction (EF ≥ 45%) and type 2 diabetes mellitus who receive treatment with glucagon-like peptide-1 (GLP-1) receptor agonists
  Interventions: Drug: Tirzepatide (Mounjaro); Drug: dapagliflozin, empagliflozin, metformin

INTERVENTIONS:
Drug: Tirzepatide (Mounjaro) — Tirzepatide is a dual GIP and GLP-1 receptor agonist administered by subcutaneous injection once weekly. It is used to improve cardiac function and metabolic control in patients with chronic heart failure with preserved ejection fraction. Dosage and treatment duration are defined by the study protocol.
  Other Names: Dual GIP/GLP-1 receptor agonist
Drug: dapagliflozin, empagliflozin, metformin — Standard treatment according to current clinical guidelines for chronic heart failure, which may include ACE inhibitors, beta-blockers, diuretics, insulin or oral hypoglycemics as appropriate.
  Other Names: Forxiga; Jardiance; Siofor

SUMMARY:
This clinical study aims to improve the diagnosis and treatment of cardiovascular diseases in Kazakhstan by Implementing Metabolic Correction with Glucagon-Like Peptide-1 (GLP-1). These medicines are called incretin-based therapies and include GLP-1 receptor agonists and a newer dual therapy that targets both GIP and GLP-1 receptors. Such medications have already shown benefits in lowering blood sugar, reducing body weight, improving blood pressure, and lowering the risk of serious heart complications.

Cardiovascular diseases and diabetes are among the most common health problems in Kazakhstan. Many patients remain undiagnosed or receive treatment only after their condition becomes severe. This study seeks to address these challenges by testing how well dual incretin therapy works in improving heart health, blood sugar control, and overall metabolic status in adults who have both chronic heart failure and type 2 diabetes.

Participants in the study will receive a detailed health evaluation at the beginning, including heart tests, blood work, and genomic profiling. Genomic testing will help researchers understand whether certain genetic features affect how patients respond to this therapy. After the initial assessment, participants will start treatment with a GIP/GLP-1 receptor agonist and will be monitored every few months for a total of 40 weeks. During these visits, their heart function, blood sugar levels, weight, and other health indicators will be checked to ensure both safety and effectiveness.

The main hypothesis of the study is that dual incretin therapy will improve heart function, reduce cardiometabolic risks, and show measurable benefits in patients with both chronic heart failure and type 2 diabetes. The study also assumes that a person's genetic profile may influence how well they respond to treatment.

By the end of the project, researchers hope to better understand how these medications work in the Kazakhstani population and to use these findings to support more personalized, effective, and modern approaches to treating cardiovascular diseases.

DETAILED DESCRIPTION:
Title: Improving the Diagnosis and Treatment of Cardiovascular Diseases in Kazakhstan by Implementing Metabolic Correction with Glucagon-Like Peptide-1 (GLP-1).

Overview:

Cardiovascular diseases (CVDs) remain the leading cause of morbidity and mortality worldwide and in Kazakhstan. The increasing prevalence of chronic conditions such as heart failure with preserved ejection fraction (HFpEF), obesity, and type 2 diabetes mellitus (T2DM) underscores the urgent need for integrated therapeutic approaches targeting both metabolic and cardiovascular risk factors. Despite advances in pharmacological and interventional care, standard therapies often fail to address underlying metabolic dysfunction and systemic inflammation, which are critical drivers of CVD progression.

Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) and dual incretin receptor agonists such as tirzepatide represent a novel class of therapeutics with multimodal actions. These agents improve glycemic control, promote weight loss, modulate lipid metabolism, and exert direct cardiovascular protective effects, including endothelial stabilization, reduction of oxidative stress, attenuation of systemic inflammation, and modulation of myocardial remodeling.

This study aims to improving the Diagnosis and Treatment of Cardiovascular Diseases in Kazakhstan by Implementing Metabolic Correction with Glucagon-Like Peptide-1 (GLP-1) therapies. Integration of genomic profiling seeks to identify genetic determinants of therapeutic response, enabling a precision medicine approach and supporting the development of population-specific treatment guidelines.

Scientific Rationale:

The pathophysiology of HFpEF and T2DM involves intricate mechanisms, including insulin resistance, chronic low-grade inflammation, endothelial dysfunction, myocardial stiffness, and impaired diastolic relaxation. Conventional management strategies-such as antihypertensive therapy, lipid-lowering agents, and glucose-lowering medications-primarily target downstream clinical manifestations rather than these upstream pathogenic mechanisms.

GLP-1 receptor agonists act through multiple pathways to improve cardiometabolic health:

* Pancreatic Effects: Enhance glucose-dependent insulin secretion, suppress inappropriate glucagon release, and improve postprandial glycemia.
* Gastrointestinal Effects: Delay gastric emptying and increase satiety, facilitating weight loss and improved energy balance.
* Cardiovascular Effects: Stabilize endothelial function, reduce oxidative stress, inhibit pro-inflammatory cytokines, and promote vasodilation through nitric oxide-mediated pathways.
* Metabolic Effects: Improve insulin sensitivity, reduce visceral adiposity, and positively affect lipid profiles.

Dual incretin receptor agonists, such as tirzepatide, combine GLP-1 and glucose-dependent insulinotropic polypeptide (GIP) receptor activation, synergistically enhancing insulinotropic and metabolic effects. Tirzepatide has demonstrated superior reductions in HbA1c and body weight compared with GLP-1 monotherapy in large clinical trials and is associated with emerging evidence for cardiovascular risk reduction.

Kazakhstan presents a unique population for investigating these therapies, given the rising burden of obesity, diabetes, and CVD, as well as under-characterized genetic determinants of therapeutic response. By incorporating genomic profiling, this study will elucidate population-specific factors that influence efficacy, safety, and metabolic outcomes, thereby facilitating personalized treatment strategies.

Study Design:

This is a multicenter, prospective, interventional, non-randomized clinical trial conducted at leading cardiology centers in Kazakhstan. The study duration for each participant is 40 weeks, with regular follow-up visits every 12 weeks. Adult men and women aged 18-75 years with clinically diagnosed HFpEF and T2DM are eligible for enrollment, following informed consent and confirmation of eligibility criteria.

Intervention:

Participants meeting inclusion criteria will receive dual GIP/GLP-1 receptor agonist therapy (tirzepatide) according to recommended dosing regimens. Concomitant standard-of-care cardiovascular therapy-including antihypertensive and lipid-lowering medications-will continue to ensure comprehensive management. Therapy titration will be performed according to tolerability, metabolic response, and safety monitoring.

Clinical Assessments and Monitoring:

* Cardiovascular Evaluation: Echocardiography assessing left atrial volume, E/e' ratio, left ventricular mass, and diastolic function; electrocardiography for rhythm assessment; blood pressure monitoring.
* Metabolic Assessment: Laboratory tests including HbA1c, fasting plasma glucose, lipid profile, renal and liver function tests.
* Inflammatory Biomarkers: High-sensitivity C-reactive protein (hsCRP), interleukin-6 (IL-6), NT-proBNP.
* Anthropometry: Body weight, BMI, waist-to-hip ratio, body composition analysis using bioimpedance.
* Functional Capacity: 6-minute walk test (6MWT), NYHA functional classification.
* Quality of Life Assessment: SF-36 for general physical and mental health; MLHFQ for heart failure-specific quality of life.
* Safety Monitoring: Adverse event reporting, hypoglycemia monitoring, gastrointestinal symptoms, injection site reactions, and laboratory abnormalities.

Genomic Profiling:

Peripheral blood samples will be collected at baseline for whole exome or whole genome sequencing. Bioinformatic pipelines will be applied for variant calling, annotation, and association analysis. Variants will be evaluated for associations with therapeutic efficacy, metabolic response, cardiovascular outcomes, and adverse events. Significant findings will be cross-referenced with pharmacogenomic databases to identify functionally relevant polymorphisms.

Scientific Objectives:

Primary: Evaluate changes in glycemic control (HbA1c), body weight, BMI, and echocardiographic parameters of diastolic function over 40 weeks of therapy.

Secondary: Assess improvements in functional capacity, lipid and metabolic biomarkers, inflammatory profiles, and quality of life. Monitor incidence of cardiovascular events, hospitalizations, and adverse events.

Exploratory: Identify genomic markers associated with differential response to therapy and develop predictive pharmacogenomic models to inform individualized treatment strategies.

Data Analysis Plan:

Descriptive statistics will summarize baseline demographics, clinical characteristics, and laboratory findings. Continuous variables will be expressed as mean ± SD or median (IQR), and categorical variables as frequencies and percentages. Paired t-tests or Wilcoxon signed-rank tests will assess within-group changes, while ANOVA or Kruskal-Wallis tests will evaluate subgroup differences (e.g., by genotype, sex). Multivariate regression models will adjust for confounders such as age, sex, baseline metabolic status, and concomitant medications.

Genomic analyses will integrate sequence data with clinical outcomes to identify variants associated with efficacy and safety. Multiple testing corrections and functional annotation will be applied to ensure robust findings. Data will be stored securely and analyzed using validated statistical and bioinformatic software platforms.

Expected Outcomes:

The study is anticipated to demonstrate significant improvements in glycemic control, weight reduction, and diastolic cardiac function. Anti-inflammatory and metabolic biomarker profiles are expected to improve, accompanied by enhanced quality of life and functional capacity. Genomic analysis will identify patient subgroups most responsive to therapy, enabling predictive pharmacogenomic models tailored to the Kazakh population.

Significance and Future Perspectives:

This study represents one of the first comprehensive evaluations of dual incretin therapy in Central Asia. By integrating clinical, metabolic, and genomic data, it aims to:

* Provide evidence-based guidance for the use of GLP-1 and dual incretin therapies in Kazakhstan.
* Support the development of national guidelines for HFpEF and T2DM management.
* Establish a national biobank and genomic dataset for cardiometabolic research.
* Promote precision medicine and improve long-term cardiovascular outcomes in the Kazakh population.
* Ultimately, the study addresses both local and global health priorities by advancing integrated, individualized care for patients with cardiometabolic disease and demonstrating a model for translational research in emerging healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with preserved ejection fraction (left ventricular ejection fraction not ≤ 45%)
* Type 2 diabetes mellitus (T2DM) with HbA1c level between ≥7.0% and ≤10.5%
* Ongoing treatment for T2DM (e.g., metformin and/or sulfonylureas, or basal insulin therapy)
* Stable body weight (±5%) for at least 3 months prior to screening
* Body mass index (BMI) ≥ 25 kg/m²
* Possible inclusion of patients with chronic pancreatitis in remission
* Aged 18 years or older, and not older than 75 years
* Both male and female participants

Exclusion Criteria:

* Type 1 diabetes mellitus
* Exacerbation of chronic pancreatitis
* Acute pancreatitis
* Proliferative diabetic retinopathy, diabetic maculopathy, or non-proliferative diabetic retinopathy
* History of bariatric (weight-loss) surgery or conditions associated with delayed gastric emptying
* Acute or chronic hepatitis
* Chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73 m²
* Myocardial infarction or stroke within the past 2 months
* Medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2) in the participant or a first-degree relative
* Use of any other antidiabetic medications (except metformin and/or sulfonylureas and basal insulin) within the past 3 months
* Use of weight loss medications, including over-the-counter drugs, within the past 3 months
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorders within the past 2 years
* Healthy individuals (no cardiovascular or metabolic disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP levels from baseline to Week 24 | Baseline to Week 24
  N-terminal pro-B-type natriuretic peptide (NT-proBNP) is a biomarker of heart failure severity. A reduction in NT-proBNP reflects improved cardiac function. This outcome assesses the effect of tirzepatide on heart failure status.

SECONDARY OUTCOMES:
Changes in clinical parameters associated with heart failure and type 2 diabetes mellitus | Baseline to Week 24
  Change in body weight (kg)
Changes in metabolic associated with type 2 diabetes mellitus | Baseline to Week 24
  Change in HbA1c (%)
Assessment of the Overall Condition of Patients Before and After the Study | Baseline to Week 40
  - Changes in clinical parameters associated with heart failure, including quality-of-life assessment using the SF-36 questionnaire for general physical and mental health and the Minnesota Living with Heart Failure Questionnaire (MLHFQ) for heart failure-specific quality of life.
  This parameter will be assessed individually, twice during the study period: at baseline and at the end at week 40 of the study, to assess the overall metabolic and cardiac impact of tirzepatide in patients with heart failure with preserved ejection fraction and type 2 diabetes mellitus.
Changes clinical parameters associated with heart failure | Baseline to Week 32
  -Change in left ventricular ejection fraction (LVEF) by echocardiography
Changes in clinical parameters associated with heart failure and type 2 diabetes mellitus | Baseline to Week 24
  Height parameters (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- PI "National Laboratory Astana", Nazarbayev University, Astana, Kazakhstan, Kazakhstan

DOCUMENTS (1):
  • Informed Consent Form (2025-12-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT07303556/ICF_001.pdf